CLINICAL TRIAL: NCT06410872
Title: Risk Taking and Decision-making in Cluster Headache Patients
Acronym: RiCH
Status: Completed | Type: Observational
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, RolfFronczek, MD, PhD, Leiden University Medical Center
Other Study IDs: NL68327
Record Dates: First submitted 2019-10-08; First posted 2024-05-13 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Cluster Headache
MeSH Terms: conditions — Cluster Headache

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Episodic cluster headache: Patients diagnosed according to ICHD3 criteria with episodic cluster headache
  Interventions: Diagnostic Test: BART Task
- Chronic cluster headache: Patients diagnosed according to ICHD3 criteria with chroniccluster headache
  Interventions: Diagnostic Test: BART Task
- Migraine: Patients diagnosed according to ICHD3 criteria with migraine (MA and MO)
  Interventions: Diagnostic Test: BART Task
- Healthy controls: Healthy controls, sex- and age-matched without current diagnosis of headache disorder
  Interventions: Diagnostic Test: BART Task

INTERVENTIONS:
Diagnostic Test: BART Task — The Zuckerman's Sensation Seeking Scale version-V (SSS-V) - Four-factor score, The Barret Impulsiveness Scale (BIS), Gormally's Binge Eating Scale (BES), The World Health Organization-developed AUDIT (Alcohol Use Disorders Identification Test) screen, The CAGE questionnaire for substance abuse-adapted to include drugs, Gamblers Anonymous's 20 Questions (GA20), Hospital Anxiety and Depression Scale (HADS)
  Other Names: Questionnaires

SUMMARY:
Since there is conflicting and insufficient data regarding CH personality and addictive behaviour, the investigators will investigate risk- and reward seeking behaviour in people with cluster headache. If an increased tendency towards this behaviour is shown, it will add to the clinical knowledge of cluster headache and possible lead to insights in a common biological susceptibility.

DETAILED DESCRIPTION:
Cluster headache is a severe primary headache disorder. In clinical anecdotes, people with cluster headache frequently report use of tobacco and illicit drugs. Furthermore, addictive behaviours and tattoos are considered to be more common in people with cluster headache than in the general population. The causality of these associations remains unclear. A common biological susceptibility has been proposed, predisposing people to both addictive behaviour and cluster headache. On the other hand, a role of illicit drug exposure in cluster headache pathophysiology has been suggested. The increased use of tobacco and illicit drugs could also reflect attempts to treat cluster headache attacks. In this explorative study the investigators will assess both subjective and objective measures reflecting addictive behaviour and risk- and reward seeking in cluster headache. This will add to the clinical knowledge of cluster headache and possible lead to insights in a common biological susceptibility.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-64 years
* Normal or corrected vision with acuity up to 20/60
* Presence of episodic (n=35) or chronic (n=35) cluster headache or migraine with or without arua (n=35), diagnosed according to the International Classification of Headache Disorders criteria, 3rd edition (ICHD-3, 3.1.1)

Exclusion Criteria:

* Diagnosis of uncorrected visual problems (myopia/presbiopia, peripheral vision problems or legal blindness)
* Current diagnosis of generalized anxiety disorder, depression or other psychiatric illness
* Other acute, unstable medical conditions or serious chronic diagnoses

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People with episodic (n=35) and chronic cluster headache (n=35) will be recruited from the Neurology outpatient clinic of Leiden University Medical Centre. Migraineurs (n=35) will be recruited from the LUMINA pool from people with migraine who have previously expressed interest in being contacted for future studies. Healthy controls (n=35) will be recruited from a pool of prior research-study participants, who have previously expressed interest in being contacted for future studies. We aim to achieve a 3:1 male:female ratio.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2019-04-23 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Difference in mean total score on the Zuckerman Sensation Seeking Scale between groups | One time-point
  Between group difference
Difference in mean total number of pumps during second trial between groups | One time-point
  Between group difference

SECONDARY OUTCOMES:
Difference in mean scores on the array of psychometric tests between groups | One time-point
  Between group difference
Difference in mean scores on the BART between groups and between the first and second BART within groups | One time-point
  Average # of pumps, Exploded Balloons

CONTACTS AND LOCATIONS:
Overall Officials: Rolf Fronczek, MD / PhD, Principal Investigator — Neurologist LUMC
Locations (1):
- LUMC, Leiden, South Holland, Netherlands